CLINICAL TRIAL: NCT06682117
Title: A Clinical Study of Personalized Self-DC Vaccine Targeting Neoantigen in Treatment of Advanced Solid Tumor
Acronym: Neo-DCV-001
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ji Dongmei, associate professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neo-DCV-001
Record Dates: First submitted 2024-09-19; First posted 2024-11-12 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Treatment; Neoantigen; Vaccine; Solid Tumor Cancer
Keywords: advanced solid tumors; DC vaccine; neoantigen
MeSH Terms: interventions — lentiviral minigene vaccine of COVID-19 coronavirus

STUDY DESIGN:
Intervention Model Description: This is a single arm, single center, open label study designed as "3+3" model to explore the MTD and DLT of personalized self-DC vaccine targeting neoantigen in treatment of advanced solid tumor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): Patients will received DC vaccine infusions.
  Interventions: Drug: DC Vaccine

INTERVENTIONS:
Drug: DC Vaccine — Patients will receive Neo-DC vaccine infusion either by dose 1 (1×10^7 cells/time) or dose 2 (5×10^7 cells/time) every 7 days, four cell infusions are one treatment cycle.
  The dose limited toxity observation time is within 28 days after the first Neo-DC vaccine infusion.
  If the efficacy is evaluated as clinical benefit (CR/PR/SD) or immune unconfirmed progress ( iUPD), treatment cycle can be continued until the completion of four Neo-DC vaccine administrations or disease progression (iCPD by iRECIST) or start new anti-tumor treatment or stop treatment by other reasons.

SUMMARY:
This is a clinical study of personalized self-DC vaccine targeting neo-antigen (Neo-DC vaccine) in the treatment of advanced solid tumors.

DETAILED DESCRIPTION:
This is a clinical study of personalized self-DC vaccine targeting neo-antigen (Neo-DC vaccine) in the treatment of advanced solid tumors (especially head and neck cancer, non-driver gene sensitive mutation of non-small cell lung cancer). The investigators plan to enroll about 9 patients to explore the dose limited toxicity or recommended dose for future study of Neo-DC vaccine. The study is designed as 3 plus 3 model, and set two dose levels.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years.
2. Histologically or cytologically confirmed advanced solid tumor, with at least one tumor lesion measurable (basis RECIST1.1 standard).
3. HLA typing was HLA-A0201/1101/2402 (containing at least one of the typing, according to the central laboratory issued).
4. Paraffin-embedded tumor tissue sections or biopsy tumor tissues within 3 years (for tumors with easy sampling).
5. Before enrollment, systemic standard treatment failure or standard treatment intolerance, and meet the following tumor requirements : new antigen positive（head and neck tumors, non-small cell lung cancer without driver genes (no EGFR sensitive mutation / ALK fusion positive), esophageal squamous cell carcinoma).
6. Voluntary to participate in clinical research ; the person or legal guardian fully understands and is informed of this study and sign the informed consent; willing to follow and be able to complete all test procedures;
7. ECOG score 0-1.
8. Have a venous access to meet single collection or venous blood collection;
9. Expected survival time ≥ 6 months.
10. Subjects were willing to study the use of reliable contraceptive methods during treatment and within 3 months after the end of treatment, and women of childbearing age.
11. Have adequent organ functions.
12. Before administration of Neo-DCV injection : 1) any chemotherapy, targeted drugs, immune checkpoint inhibitors, other clinical trial research drugs, traditional Chinese medicine with anti-tumor indications and other anti-tumor treatments received have passed the 4-week elution period, and the toxic and side effects returned to grade 1 or lower (except for alopecia, vitiligo and other tolerable events judged by researchers) ; 2) If undergoing major surgery within 3 weeks, the adverse reactions have returned to grade 1 or lower.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with a history of severe immediate allergies to the cells and any drugs used in this study.
3. Those with a history of organ transplantation.
4. Known central nervous system metastasis.
5. Any active autoimmune disease or any autoimmune disease that has been determined by the researchers to be unsuitable for this study.
6. Uncontrolled concomitant diseases or infectious diseases, such as the need for systemic antibiotics within 2 weeks before enrollment.
7. Suffering from severe liver and kidney function damage (liver, kidney treatment but still not controllable, biochemical indicators can not meet the inclusion criteria of NO.11, or can not control the diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease, or poor drug control of hypertension ( systolic blood pressure more than 160mmHg and/or diastolic blood pressure more than 90mmHg), or with clinical Bed meaning (e.g. activity ) of cardiovascular and cerebrovascular diseases, such as cerebrovascular accident (6 months before signing informed consent) unstable angina, myocardial infarction (within 6 months before signing informed consent), unstable angina, New York Heart Association, or any circumstances which, in the opinion of the researcher, may increase the risk of the subject or interfere with the results of the test.
8. Subjects planned to receive sugar within 4 weeks before the first Neo-DCV injection and during the study period due to certain conditions.

   Corticosteroids (prednisone or the same drug dose less than 10mg/day ) or other immunosuppressive agents were excluded.
9. Subjects were scheduled to receive Neo-DCV injection within 4 weeks before the first administration and during the study period due to certain conditions.
10. The researchers assessed that the subjects were unable or unwilling to comply with the requirements of the study protocol.
11. The defects of antigen presentation, antigen recognition and cell killing related genes were detected by sequencing.
12. There was a history of other malignant tumors in the past 5 years, except for curable basal cell carcinoma, papillary thyroid carcinoma, and uterus.
13. Subjects have any disease or medical condition that may affect the evaluation of the safety or efficacy of the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Within 28 days after the first Neo-DC vaccine cell infusion
  The incidence and severity of adverse events

SECONDARY OUTCOMES:
Objective response rate (ORR) | up 2 years
  The partial remission (PR) and complete remission rate (CR)
Dose limited toxicity | Within 28 days after the first Neo-DC vaccine cell infusion
  Dose limited toxicity within 28 days after the first Neo-DC vaccine cell infusion

OTHER OUTCOMES:
IFN-γ activity detected by ELISPOT, cell factor and T cell subsets detection. | up 2 years
  IFN-γ activity detected by ELISPOT, cell factor detected by ELISA, and T cell subsets detection by flow cytometry.
iDCR | up 2 years
  iDCR by iRECIST
iPFS | up 2 years
  iPFS by iRECIST
iDOR | up 2 years
  iDOR by iRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Xianghua Wu, M.D, Principal Investigator — Fudan University; Qinghai Ji, M.D, Principal Investigator — Fudan University; Dongmei Ji, M.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No